CLINICAL TRIAL: NCT06021171
Title: Improving the Iron Status of Athletes With Pre-, Pro- and Synbiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College (Other)
Responsible Party: Principal Investigator, Diane DellaValle, PhD, RDN, LDN, Associate Professor, Research Dietitian, King's College
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-44-0701
Record Dates: First submitted 2021-06-25; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Iron Deficiency (Without Anemia)
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled crossover trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Volunteers will be asked to mix the powder packet (e.g. supplemental functional fiber source or placebo), with any food or beverage once daily. All 3 powders are identically packaged and only visible as white powder, and all 3 powders are colorless, odorless and tasteless when mixed in a liquid or semi-solid food. Instructions and education to both groups will be identical. Packets were sent to the Researcher pre-packaged and pre-labeled as A, B, C by the product company.
  Subject randomization to treatment order was completed using random number generator by a Research Assistant not involved in direct contact with subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular Girl (Sunfiber + Bifidobacterium lactis) (Active Comparator): Regular Girl, a synbiotic supplement containing the Prebiotic Sunfiber + Bifidobacterium Lactis
  Interventions: Dietary Supplement: Partially hydrolyzed guar gum + bifidobacterium lactis
- Maltodextrin (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin
- Sunfiber (Active Comparator): SunFiber, a prebiotic fiber supplement
  Interventions: Dietary Supplement: Partially hydrolyzed guar gum

INTERVENTIONS:
Dietary Supplement: Partially hydrolyzed guar gum + bifidobacterium lactis — Synbiotic Supplement: Contains 5 grams of prebiotic fiber (Sunfiber®) and 8 billion active probiotics (Bifidobacterium lactis).
  Other Names: RegularGirl
  Arms: Regular Girl (Sunfiber + Bifidobacterium lactis)
Dietary Supplement: Partially hydrolyzed guar gum — 5 g Partially hydrolyzed guar gum
  Other Names: SunFiber
  Arms: Sunfiber
Dietary Supplement: Maltodextrin — 5 g Maltodextrin
  Arms: Maltodextrin

SUMMARY:
Iron deficiency (ID) is the most common micronutrient deficiency worldwide, and poor iron bioavailability is a major cause. While 30% of female athletes are affected by ID, and its consequences are highly relevant to athletic performance, ID affects women and children around the world with consequences just as relevant, if not more so (e.g. school performance, work capacity and thus wage earning). With poor iron absorption being a cause of ID in active women, it is especially important to discover simple ways to improve iron (Fe) uptake. While some studies have suggested that consumption of prebiotic fiber may improve Fe absorption in animal models, there have been few studies examining the effects of synbiotic supplementation (consumption of both a prebiotic and probiotic that work together) on Fe uptake in adult females (athletes and non-athletes).

A recent pilot study demonstrated a substantial improvement in Fe uptake in female athletes after 4 and 8 weeks of synbiotic supplementation compared to placebo during Fe repletion with a low dose of ferrous sulfate (FeSO4). If synbiotic supplementation can improve the Fe bioavailability of FeSO4 (which is ~30%) in ID women during repletion of Fe status, it could possibly improve the Fe bioavailability of non-heme Fe sources, as well as mixed meals.

Research Question: What is the effect of synbiotic supplementation (a supplement containing a prebiotic + a probiotic), compared to prebiotic supplementation or a placebo, on Fe uptake and the gut microbiome in ID athletes during low-dose Fe repletion?

Hypothesis: In the proposed study, we hypothesize that synbiotic supplementation along with Fe repletion with a low dose of FeSO4 will have greatest impact on athletes' Fe uptake due to alterations in the microbiome, which will be assessed.

DETAILED DESCRIPTION:
The following Specific Aims will help us to answer this research question: To screen the iron status of athletes at the beginning of training season and determine the prevalence of anemia and iron depletion on our NCAA Division III campus. To determine the differences in Fe uptake with consumption of a synbiotic, prebiotic, and placebo supplements along with low-dose Fe supplementation in ID athletes. To determine the differences in the microbiome with consumption of a synbiotic, prebiotic, and placebo supplements along with low-dose Fe supplementation in ID female athletes. This aim will help us mechanism behind change in iron status with a functional fiber (e.g. synbiotic supplementation).

This data is essential to advance our understanding of how Fe uptake in active persons can be enhanced by functional fiber supplementation, as well as by REAL foods containing functional fibers, which could help ameliorate ID not only for athletes here in the US but for people around the globe.

The design is a randomized, placebo-controlled crossover trial, which will use each participant as her/his own control, in addition to a placebo treatment being administered in a counter-balanced order with the other treatments.

Participants: King's is a Division III College and currently has >85 eligible female athletes on the rosters of a variety of competitive sports teams. During a recent RCT, about 30 active women were screened and >30% were ID (1). For the proposed study, given the effect size observed in previous work (6), we need n=10 to complete the 18-week randomized crossover trial (e.g. so recruiting n=13 would allow for a "normal" 20% attrition rate during the trial due to injuries, illnesses, etc).

Iron Status Screening: Athletes from King's will be asked to volunteer via recruitment email. To address Aim 1, at baseline (and after NCAA health clearance), athletes will have their iron status screened via venous blood sample at the beginning of their season in the Human Performance Lab in the Alley Center (Complete Blood Count, which includes Hgb); Serum ferritin; C-Reactive Protein for inflammation adjustment of ferritin). Anthropometrics and body composition will be measured and health, dietary and training information will also be collected. Standard demographic information, and medical history will be self-reported by each participant using computer-based questionnaires. All athletes with normal iron status (Hgb >12.0 g/dL AND sFer>30.0 µg/L) will be given their iron status results and offered a Nutrition Consultation by a MS Nutrition Student under the supervision of the PI. Athletes will not be eligible to participate in the study if pregnant, wishing to become pregnant, breastfeeding, having a condition or taking medication impacting Fe status, or not healthy enough to train/participate in their sport.

Crossover Trial: To address Aims 2 and 3, women athletes identified as ID (sFer<30.0 µg/L) will be invited to participate in a 18-week double-blind, randomized, crossover trial with concurrent daily Fe supplementation (100 mg FeSO4/d, Puritan's Pride). Participating ID athletes will receive the following treatments for 4 weeks each, in a randomized, counter-balanced order: a) synbiotic supplement (RegularGirl), b) prebiotic supplement (SunFiber), and c) placebo (maltodextrin). There will be a 3-week wash-out period between treatments (see Figure 1). In our pilot study, we observed a strong response within a 4-week time period.

Volunteers will be asked to mix the supplemental functional fiber source (or placebo) packet, all identically packaged and only visible as white powder, with any food or beverage once daily. They will also asked to consume 100 mg FeSO4 per day as a single low-dose Fe tablet once per day, either in the morning or in the evening, avoiding consumption with coffee/tea or supplemental calcium source. Throughout the 18-week study, athletes will be asked to complete a daily training, medication, compliance, stool (using the Bristol Stool Scale, BSS) and GI symptom log. Compliance will also be measured by research staff via weekly pill and packet counts.

Iron status (as described in Screening above) and dietary intake (via 24-h recall and FFQ) will be measured at the beginning and end of each treatment point of the trial (see "X" in Figure 1). Fecal samples will be collected at beginning and end of each timepoint for analysis of the microbiome (see "X" in Figure 1) using self-collection vials provided (OMNIgene-GUT, OMG-200, DNA GenoTek). Volunteers will not be asked to alter their usual food/ dietary intake in any way during the trial. At the end of the study, athletes will be given their endpoint lab results and offered a Nutrition Consultation by a MS Nutrition Student under the supervision of the PI.

Iron status (as described in Screening above) and dietary intake (via 24-h recall and FFQ) will be measured at the beginning and end of each treatment point of the trial (see "X" in Figure 1). Fecal samples will be collected at beginning and end of each timepoint for analysis of the microbiome (see "X" in Figure 1) using self-collection vials provided (OMNIgene-GUT, OMG-200, DNA GenoTek). Volunteers will not be asked to alter their usual food/ dietary intake in any way during the trial. At the end of the study, athletes will be given their endpoint lab results and offered a Nutrition Consultation by a MS Nutrition Student under the supervision of the PI.

Time and effort: 15.5 hours over the 18 week study Blood sampling and body measurements will take about 15 min, 6x during the trial (1.5 h total) Completion of forms will take about 15 min 6 x during the trial (1.5 h total) Stool collection will take about 5 min, 6 times during trial (0.5 h total) Meeting at the Alley Center Human Performance Lab weekly will take ~ 5 min, 18x over the course of the study (1.5 h total) Consumption of iron supplement and packet every day and daily record-keeping will take <5 min/day * 126 days during 18 week study (<10.5 h total)

Data analysis plan: All analyses of sFer will be adjusted for inflammation. Briefly, GLM Repeated measures ANOVA will be used to assess the effect of the treatments on iron status, GI symptoms, etc. (Time-by-Tx effects will be examined). All statistical analyses will be performed using SPSS (most recent version), and results will be considered statistically significant at p<0.05 for main effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* currently participating in or training for their sport

Exclusion Criteria:

* Pregnant, or wishing to become pregnant
* Breastfeeding
* Having a condition or taking medication impacting iron status
* Not healthy enough to train for/participate in their sport.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Blood serum level of ferritin | baseline (0), 4, 8, 12, 16, 18 weeks
  biomarker of iron status, iron stores, use to calculate Total body iron
Blood level of hemoglobin | baseline (0), 4, 8, 12, 16, 18 weeks
  biomarker of iron status
Blood serum level of soluble transferrin receptor | baseline (0), 4, 8, 12, 16, 18 weeks
  biomarker of iron status, tissue iron status, use to calculate Total body iron
Gut microbiome data | baseline (0), 4, 8, 12, 16, 18 weeks
  Fecal samples to yield gut bacterial taxa

CONTACTS AND LOCATIONS:
Overall Officials: Diane M. DellaValle, Principal Investigator — King's College
Locations (1):
- King's College, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported, after deidentification (text, tables, figures, appendices).
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact dianedellavalle@kings.edu.

REFERENCES:
- [Background] DellaValle DM, Haas JD. Impact of iron depletion without anemia on performance in trained endurance athletes at the beginning of a training season: a study of female collegiate rowers. Int J Sport Nutr Exerc Metab. 2011 Dec;21(6):501-6. doi: 10.1123/ijsnem.21.6.501. PMID 22089308
- [Background] Dellavalle DM, Haas JD. Iron status is associated with endurance performance and training in female rowers. Med Sci Sports Exerc. 2012 Aug;44(8):1552-9. doi: 10.1249/MSS.0b013e3182517ceb. PMID 22382172
- [Background] Sandroni A, House E, Howard L, DellaValle DM. Synbiotic Supplementation Improves Response to Iron Supplementation in Female Athletes during Training. J Diet Suppl. 2022;19(3):366-380. doi: 10.1080/19390211.2021.1887423. Epub 2021 Feb 22. PMID 33615951
- [Background] DellaValle DM, Glahn RP, Shaff JE, O'Brien KO. Iron Absorption from an Intrinsically Labeled Lentil Meal Is Low but Upregulated in Women with Poor Iron Status. J Nutr. 2015 Oct;145(10):2253-7. doi: 10.3945/jn.115.217273. Epub 2015 Sep 2. PMID 26338889
- [Background] Scholz-Ahrens KE, Schrezenmeir J. Inulin and oligofructose and mineral metabolism: the evidence from animal trials. J Nutr. 2007 Nov;137(11 Suppl):2513S-2523S. doi: 10.1093/jn/137.11.2513S. PMID 17951495
- [Background] Freitas Kde C, Amancio OM, de Morais MB. High-performance inulin and oligofructose prebiotics increase the intestinal absorption of iron in rats with iron deficiency anaemia during the growth phase. Br J Nutr. 2012 Sep 28;108(6):1008-16. doi: 10.1017/S0007114511006301. Epub 2011 Dec 15. PMID 22172251
- [Background] Laparra JM, Diez-Municio M, Herrero M, Moreno FJ. Structural differences of prebiotic oligosaccharides influence their capability to enhance iron absorption in deficient rats. Food Funct. 2014 Oct;5(10):2430-7. doi: 10.1039/c4fo00504j. Epub 2014 Aug 11. PMID 25109275
- See also: Website for RegularGirl Product — https://regulargirl.com/products/copy-of-regular-girl-on-the-go
- See also: Website for SunFiber Product — https://sunfiber.com/products/